CLINICAL TRIAL: NCT01888003
Title: The Benefits of a Preoperative Anemia Management Program
Acronym: PAMP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Thomas R. Vetter, MD, MPH, Maurice S. Albin Professor of Anesthesiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F130117001
Record Dates: First submitted 2013-03-20; First posted 2013-06-27 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Anemia, Iron-Deficiency
Keywords: anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — Ferric Oxide, Saccharated; Epoetin Alfa; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anemia Treatment Group (AMG) (Active Comparator): Group of patients who are diagnosed preoperatively as being anemic (defined as a Hgb < 13.0 g/dL and MCV < 100 fL, with a hematocrit between 30% and 39%, for males and females), who will receive an ESA (PROCRIT) and iron (Venofer) preoperatively.
  Interventions: Drug: Iron sucrose; Drug: Epoetin Alfa; Other: Blood Transfusion
- Conventional Treatment Group (CTG) (Other): Group of patients who are diagnosed preoperatively as being anemic (defined as a Hgb < 13.0 g/dL and MCV < 100 fL, with a hematocrit between 30% and 39%, for males and females), who will receive our current, conventional perioperative standard of care, which does not involve any preoperative anemia management (other than laboratory testing). CTG patients will undergo routine perioperative laboratory testing/screening.
  Interventions: Other: Blood Transfusion
- Non Anemia Group (NAG) (Other): Group of patients who are not anemic preoperatively, who will receive our current, conventional perioperative standard of care.
  Interventions: Other: Blood Transfusion

INTERVENTIONS:
Drug: Iron sucrose — AMG patients will receive a standardized and well-accepted intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days and -7 days before their planned surgery, and if indicated, based upon laboratory testing on the day of their surgery (if patient has a Hgb < 13.0 g/dL and hematocrit between 30% and 39%, for males and females). An additional dose will be given on postoperative day 2.
  Other Names: (Venofer®)
  Arms: Anemia Treatment Group (AMG)
Drug: Epoetin Alfa — AMG patients will receive a standardized and well-accepted subcutaneous dose of 40,000 IU of epoetin alfa (PROCRIT®) plus an intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days and -7 days before their planned surgery, and if indicated, based upon laboratory testing on the day of their surgery (if patient has a Hgb < 13.0 g/dL and hematocrit between 30% and 39%, for males and females).
  Other Names: PROCRIT®
  Arms: Anemia Treatment Group (AMG)
Other: Blood Transfusion — An evidence-based, goal-directed blood transfusion protocol will be applied in AMG, CTG, and NAG patients during and after their surgical procedure to control for health provider variation in transfusion criteria and practices. This blood conservation protocol will consist primarily of the application of a restrictive transfusion trigger (Hgb < 8 g/dl) (21,22) but will also take into consideration the patient's intraoperative estimated allowable blood loss and hemodynamic stability.

SUMMARY:
The goal of this study is to gain further insight into the comparative effectiveness of treating patients, who are found to be anemic before their elective surgery, with a series of weekly subcutaneous doses of a drug given before surgery, which stimulates the natural production of red blood cells (a so-called erythropoietic stimulating agent [ESA]) along with intravenous iron, in reducing the need for blood transfusions (donated by someone other than the patient) during and after adult total hip arthroplasty (hip replacement surgery). The effects of a Preoperative Anemia Management Program (PAMP) on the patient's quality of recovery, health-related quality of life, fatigue, and rehabilitation pattern after surgery will also be examined. A cost-effectiveness analysis will be performed to compare the cost of these commercially available, FDA-approved medications versus the cost of transfused blood

DETAILED DESCRIPTION:
Patient blood management (PBM) involves the timely and conscientious use of the current best evidence in making medical and surgical decisions about the care of patients to maintain red blood cell levels, optimize blood clotting, and minimize blood loss, in an effort to improve patient outcome. PBM focuses on the treatment of the individual patient and comprises transfusion therapy and drug therapy. PBM is based on three points: (1) optimization of the (preoperative) red blood cell volume, (2) reduction of diagnostic, therapeutic, or intraoperative blood loss, and (3) increasing individual tolerance towards anemia and accurate blood transfusion triggers. PBM primarily identifies patients at risk for transfusion and provides a management plan aimed at reducing or eliminating anemia and the need for blood transfusion donated from someone other than the patient (allogeneic transfusion), thus reducing the risks, blood bank inventory pressures, and the escalating costs associated with transfusion. The implementation of a formal UAB Preoperative Anemia Management Program (PAMP) may help achieve consistent PBM.

Efforts will be made to coordinate patients' scheduled surgery date and their initial evaluation in the UAB Highlands Hospital Preoperative Assessment, Consultation, and Treatment (HPACT) Clinic, so that their first PACT Clinic visit occurs approximately 14 days prior to the planned total hip replacement or total knee replacement

ELIGIBILITY:
Inclusion Criteria:

1. 19 years to 80 years of age
2. American Society of Anesthesiologists 1-3 status
3. Undergoing total hip arthroplasty for osteoarthritis, (either a primary or replacement procedure, but not a revision procedure) OR avascular necrosis (AVN); OR undergoing total knee arthroplasty (replacement) for osteoarthritis

Exclusion Criteria:

1. American Society of Anesthesiologists 4 status
2. Severe anemia, defined as a hematocrit of < 30%
3. History of hypercoagulability or thrombophilia (e.g, factor V Leiden)
4. History of deep venous thrombosis (DVT) or venous thromboembolism (VTE) within last 12 months
5. Current use of anticoagulants (e.g., heparin, warfarin, dabigatran, etc)
6. Diagnosis of chronic renal insufficiency requiring dialysis
7. Morbid obesity (BMI > 40)
8. History of allergic reaction to intravenous iron
9. History of allergic reaction to an erythropoietic stimulating agent (ESA)
10. History of sickle cell disease
11. History of hemochromatosis
12. History of liver dysfunction or congestive heart failure
13. History of substance abuse disorder
14. History of major psychiatric disorder (e.g., major depression, bipolar disorder, axis II personality disorder, schizophrenia)
15. Uncontrolled hypertension (defined as a systolic pressure ≥ 160 mmHg and/or a diastolic pressure ≥ 110 mmHg)
16. History of uncontrolled cardiac arrhythmias, cerebrovascular accident (CVA), transient ischemic attack (TIA), acute coronary syndrome (ACS), or other arterial thrombosis. ACS includes unstable angina, Q wave myocardial infarction (QwMI), and non-Q wave myocardial infarction (NQMI) within 6 months
17. History of pure red cell aplasia (PRCA) after treatment with an ESA
18. History of seizure disorder
19. Any active/current cancer within the last 12 months (not including non-melanoma skin cancer)
20. Pregnancy or lactation
21. Non-native English speaker (because validated Spanish language versions of two of the patient questionnaires are not available)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Vetter, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Highlands Hospital, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anemia Treatment Group (AMG): Group of patients who are diagnosed preoperatively as being anemic (defined as a Hgb < 13.0 g/dL and MCV < 100 fL, with a hematocrit between 30% and 39%, for males and females), who will receive an ESA (PROCRIT) and iron (Venofer) preoperatively.
  Iron sucrose: AMG patients will receive a standardized and well-accepted intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days and -7 days before their planned surgery, and if indicated, based upon laboratory testing on the day of their surgery (if patient has a Hgb < 13.0 g/dL and hematocrit between 30% and 39%, for males and females). An additional dose will be given on postoperative day 2.
  Epoetin Alfa: AMG patients will receive a standardized and well-accepted subcutaneous dose of 40,000 IU of epoetin alfa (PROCRIT®) plus an intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days and -7 days before their planned surgery, and if indicated, based upon laboratory testing on the day of their surgery (if patient has
Period: Overall Study
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Started | 5 | 6 | 40
Completed | 0 | 0 | 0
Not Completed | 5 | 6 | 40
Not completed — Study Terminated | 5 | 6 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG) | Total
Number analyzed (Participants) | 5 | 6 | 40 | 51
Age, Continuous [Mean (Full Range); unit: Years] | 63 [49 to 71] | 62 [42 to 76] | 62 [44 to 79] | 62 [42 to 79]
Sex/Gender, Customized [Number; unit: participants]
  Males | 4 | 0 | 25 | 29
  Females | 1 | 6 | 15 | 22
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 40 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Requiring at Least One Blood Transfusion During Surgery.
Description: The number of subjects who had blood transfusions (at least 1) during surgery
Time Frame: During surgery (less than 1 day)
Measure: Number; unit: Participants
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Number analyzed (Participants) | 5 | 6 | 40
Participants | 0 | 0 | 0

2. Secondary Outcome: Health-related Quality of Life
Description: Health-related quality of life measured with the SF-12V2; Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Questionnaire; Oxford Hip Score or Oxford Knee Score; and Multidimensional Assessment of Fatigue (MAF) Scale
Time Frame: Baseline at 14 days before, on hospital discharge, and at two-weeks, 30 days, 60 days and 90 days after surgery
Population: No subject data was analyzed.
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Blood Transfusions After Surgery and Prior to Discharge From Hospital
Description: Number of subjects that had at least 1 blood transfusion from the end of surgery until discharge from hospital
Time Frame: post surgery through discharge, an average of 2 days
Measure: Number; unit: participants
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Number analyzed (Participants) | 5 | 6 | 40
participants | 0 | 1 | 0

4. Primary Outcome: Number of Subjects Requiring Blood Transfusions Post Hospital Discharge Through 90 Days After Surgery
Description: number of subjects requiring blood transfusions after hospital discharge through 90 days after surgery
Time Frame: post hospital discharge through 90 days after surgery
Population: Subjects dropped out of study prior to day 90
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Anemia Treatment Group (AMG): Patients diagnosed preoperatively as being anemic (defined as a Hgb < 13.0 g/dL and MCV < 100 fL, with a hematocrit between 30% and 39%, for males and females), who will receive an ESA (PROCRIT) and iron (Venofer) preoperatively.
  Iron sucrose: AMG patients will receive a standardized and well-accepted intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days and -7 days before their planned surgery, and if indicated, based upon laboratory testing on the day of their surgery (if patient has a Hgb < 13.0 g/dL and hematocrit between 30% and 39%, for males and females). An additional dose will be given on postoperative day 2.
  Epoetin Alfa: AMG patients will receive a standardized and well-accepted subcutaneous dose of 40,000 IU of epoetin alfa (PROCRIT®) plus an intravenous dose of 200 mg of iron sucrose (Venofer®) at -14 days, -7 days before their planned surgery, and if indicated, based on labs, testing on the day of their surgery
Arm/Group | Anemia Treatment Group (AMG) | Conventional Treatment Group (CTG) | Non Anemia Group (NAG)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/40
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes